CLINICAL TRIAL: NCT05269719
Title: Epidemiology of Digital Nerve Injuries in the Stockholm County
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Cecilia Mellstrand Navarro, Principal Investigator, Karolinska Institutet
Other Study IDs: Digital nerve injury, epi
Record Dates: First submitted 2021-10-07; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Digital Nerve Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Digital nerve injury, surgical treatment, isolated injury: Patient over the age of 18 with an isolated injury to a digital nerve.
  Interventions: Procedure: Suture of digital nerve
- Digital nerve injury, surgical treatment, concomittant flexor tendon injury: Patient over the age of 18 with an injury to a digital nerve and a concomittant flexor tendon injury.
  Interventions: Procedure: Suture of digital nerve

INTERVENTIONS:
Procedure: Suture of digital nerve — The digital nerves were sutured according to the discretion of the treating surgeon and the standard procedure was three epineural sutures 8.0 or 9.0 nylon under loop magnification. Concomitant tendon injuries were also sutured according to the discretion of the treating surgeon, most commonly with two loop sutures (four strand core) and a peritendinous PDS suture.

SUMMARY:
This is a registry and medical record based epidemiological description of patients with digitial nerve injuies in the Stockholm County, Sweden

DETAILED DESCRIPTION:
The primary aim of this study was to describe the epidemiology of patients with surgically repaired digital nerve injuries in a Swedish population during the period 2012 to 2018. Secondary aims included a description of the patient population, surgical treatment and rehabilitation regimens following digital nerve injury. Comparisons were made between groups consisting in patients with isolated nerve injuries and those with a concomitant flexor tendon injury.

METHODS

Patients In this cohort study, all patients treated with surgical repair of a digital nerve injury at the Department of Hand Surgery at Södersjukhuset, Stockholm, Sweden were included. Inclusion period was between 2012-01-01 and 2018-12-31. Patients were identified through the Swedish national quality registry for Hand surgery (HAKIR). Inclusion criteria were the diagnostic codes (ICD-10) for a digital nerve injury in the thumb (S64.3) or finger (S64.4) in combination with the surgical code (KKÅ97) Nomesco classification of surgical procedures for nerve repair (ACB29). A total of 1,329 patients were identified. Exclusion criteria were concomitant skeletal injury, amputations, severe soft tissue injuries, or if the injury needed microvascular reconstruction. Patients reciding outside the Stockholm region and children below 18 years of age were also excluded. A total of 1,004 patients were included for the final analysis. The study population was thereafter divided into two groups: patients with an isolated digital nerve injury and patients with a ditial nerve injry with a concomitant tendon injury. All clinical data was collected through search of medical records.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic codes (ICD-10) for a digital nerve injury in the thumb (S64.3) or finger (S64.4) in combination with the surgical code (KKÅ97) Nomesco classification of surgical procedures for nerve repair (ACB29).

Exclusion Criteria:

* concomitant skeletal injury
* amputations
* severe soft tissue injuries
* injury needed microvascular reconstruction.
* Patients reciding outside the Stockholm region and
* patient age below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated with surgical repair of a operatively for a digital nerve injury at the Department of Hand Surgery at Södersjukhuset, Stockholm, Sweden between 2012-01-01 and 2018-12-31 were included.
Sampling Method: Non-Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence | at study inclusion
  The incidence of digital nerve injury as calculated as the numbers of treated patients divided by the population at risk

SECONDARY OUTCOMES:
Demographic features of the patient cohort | at study inclusion
  date of birth, gender, injured hand, time and date of injury and surgery. Injured nerve, injury level, injury mechanism and type of injury, total or partial nerve injury, isolated nerve injury/concomitant flexor tendon injury, and postoperative complications. Smoking status, profession, numbres of visits to health care professionals.
Health care interventions | through study completion, at an average 6 months
  time from injury to surgery, time from injury to rehabilitation, types of rehabilitation, number of visits to health care personnel, days of sick leave

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Arner, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet Södersjukhuset, Department of clinical research and education, Stockholm, Sweden